CLINICAL TRIAL: NCT01546714
Title: Sexually Transmitted Infections Among African American Women Who Have Sex With Women
Acronym: WSHP
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Mississippi Medical Center (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Dr. Christina Muzny, Assistant Professor of Medicine, University of Alabama at Birmingham
Other Study IDs: ASTDA WSHP; American STD Association (Other Grant/Funding Number: 2009283)
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Sexually Transmitted Infections
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One vaginal swab and one endocervical swab to be stored for future studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AAWSW/AAWSWM: African American Women Who Have Sex with Women/African American Women Who Have Sex with Women and Men

SUMMARY:
The purpose of this study is to determine rates of sexually transmitted infections (STIs) among African American women who have sex with women (AAWSW). In addition, the study is interested in better understanding the types of risk behaviors that place AAWSW at risk for STIs. The investigators hypothesis is that AAWSW experience high rates of STIs, similar to heterosexual African American women. Knowledge gained from this study will guide development of interventions to reduce women's risk for these types of infections and will improve how AAWSW are screened for STIs.

DETAILED DESCRIPTION:
The objectives of this study are (1) To determine the prevalence of bacterial vaginosis, trichomoniasis, Chlamydia, gonorrhea, Mycoplasma genitalium, HIV, genital herpes, and syphilis and associated risk behaviors in a cohort of African American women who have sex with women (AAWSW) in Birmingham, Alabama; (2) To compare exclusive AAWSW (during the past 12 months) to African American women who have sex with women and men (AAWSWM) in terms of socio-demographic characteristics, sexual risk behavior characteristics, and STI prevalence; and(3) To perform an exploratory prospective study of an age-matched (± 2 years) sub-group of exclusive AAWSW and AAWSWM over a 12 month time period to obtain data on differences in STI risk behaviors and STI incidence rates.

ELIGIBILITY:
Inclusion Criteria:

* Female gender, self-identification as African American
* Age of 16 years or older, self report of sexual contact (oral, vaginal, or anal) with another female within the past 12 months
* English speaking
* The ability to give written informed consent.
* For the sub-groups of women being followed prospectively, they have to have at least one active female sexual partner (AAWSW group) or at least one active female and male sexual partner (AAWSWM group) at the time of enrollment into the study.

Exclusion Criteria:

* Pregnant or nursing and the inability or unwillingness to give written informed consent.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: African American women, aged 16 years or older, living in Birmingham, Alabama
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2011-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Sexually Transmitted Infection Diagnosis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Muzny, MD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - Jefferson County Health Department, Birmingham, Alabama
  - UAB Personal Health Clinic, Birmingham, Alabama

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with investigators at the Harvard School of Public Health for secondary data analysis.

REFERENCES:
- [Background] Muzny CA, Sunesara IR, Martin DH, Mena LA. Sexually transmitted infections and risk behaviors among African American women who have sex with women: does sex with men make a difference? Sex Transm Dis. 2011 Dec;38(12):1118-25. doi: 10.1097/OLQ.0b013e31822e6179. PMID 22082722
- [Background] Muzny CA, Harbison HS, Pembleton ES, Hook EW, Austin EL. Misperceptions regarding protective barrier method use for safer sex among African-American women who have sex with women. Sex Health. 2013 May;10(2):138-41. doi: 10.1071/SH12106. PMID 23369280
- [Background] Muzny CA, Rivers CA, Mena LA, Schwebke JR. Genotypic characterization of Trichomonas vaginalis isolates among women who have sex with women in sexual partnerships. Sex Transm Dis. 2012 Jul;39(7):556-8. doi: 10.1097/OLQ.0b013e31824f1c49. PMID 22706219
- [Background] Cornelius DC, Robinson DA, Muzny CA, Mena LA, Aanensen DM, Lushbaugh WB, Meade JC. Genetic characterization of Trichomonas vaginalis isolates by use of multilocus sequence typing. J Clin Microbiol. 2012 Oct;50(10):3293-300. doi: 10.1128/JCM.00643-12. Epub 2012 Aug 1. PMID 22855512
- [Background] Muzny CA, Harbison HS, Pembleton ES, Austin EL. Sexual behaviors, perception of sexually transmitted infection risk, and practice of safe sex among southern African American women who have sex with women. Sex Transm Dis. 2013 May;40(5):395-400. doi: 10.1097/OLQ.0b013e31828caf34. PMID 23588129
- [Background] Muzny CA, Sunesara IR, Austin EL, Mena LA, Schwebke JR. Bacterial vaginosis among African American women who have sex with women. Sex Transm Dis. 2013 Sep;40(9):751-5. doi: 10.1097/OLQ.0000000000000004. PMID 23949590
- [Background] Muzny CA, Rivers CA, Parker CJ, Mena LA, Austin EL, Schwebke JR. Lack of evidence for sexual transmission of genital Candida species among women who have sex with women: a mixed methods study. Sex Transm Infect. 2014 Mar;90(2):165-70. doi: 10.1136/sextrans-2013-051361. Epub 2014 Jan 15. PMID 24431188
- [Background] Austin EL, Lindley LL, Mena LA, Crosby RA, Muzny CA. Families of choice and noncollegiate sororities and fraternities among lesbian and bisexual African-American women in a southern community: implications for sexual and reproductive health research. Sex Health. 2014 Mar;11(1):24-30. doi: 10.1071/SH13145. PMID 24438825
- [Background] Muzny CA, Kapil R, Austin EL, Brown L, Hook EW 3rd, Geisler WM. Chlamydia trachomatis infection in African American women who exclusively have sex with women. Int J STD AIDS. 2016 Oct;27(11):978-83. doi: 10.1177/0956462415604092. Epub 2015 Sep 18. PMID 26384942
- [Background] Agenor M, Austin SB, Kort D, Austin EL, Muzny CA. Sexual Orientation and Sexual and Reproductive Health among African American Sexual Minority Women in the U.S. South. Womens Health Issues. 2016 Nov-Dec;26(6):612-621. doi: 10.1016/j.whi.2016.07.004. Epub 2016 Aug 18. PMID 27546567
- [Result] Muzny CA, Austin EL, Harbison HS, Hook EW 3rd. Sexual partnership characteristics of African American women who have sex with women; impact on sexually transmitted infection risk. Sex Transm Dis. 2014 Oct;41(10):611-7. doi: 10.1097/OLQ.0000000000000194. PMID 25211257
- [Result] Muzny CA, Kapil R, Austin EL, Hook EW, Geisler WM. Lower sexually transmissible infection prevalence among lifetime exclusive women who have sex with women compared with women who have sex with women and men. Sex Health. 2014 Dec;11(6):592-3. doi: 10.1071/SH14181. PMID 25435197